CLINICAL TRIAL: NCT04460573
Title: Improving the Science of Adherence Reinforcement and Safe Mobility in People With Diabetic Foot Ulcers Using Smart Offloading
Brief Title: Smart Boot Use to Measure Offloading Adherence
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, David Armstrong, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-20-00526
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: prospective, comparative randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Reference Group (Active Comparator): The group 1 will receive above-standard of care intervention, which includes wearing a standard removable boot and enhanced eductaion with weekly adherence reinforcement. In this group, participants are interviewed weekly, adherence is reviewed, and education is reinforced at each visit. Participants are instructed to wear the offloading device at all times, including during rest and at night, and not to remove it at any time.
  Interventions: Device: Offloading Boot
- Group 2: Control Group (Active Comparator): The control group uses removable offloading and represents the standard of care. These participants receive education at baseline and are advised to wear the offloading device during walking or standing; however, they are allowed to remove it during rest and sleep.
  Interventions: Device: Offloading Boot
- Group 3: SmartBoot (Experimental): The SmartBoot group follows a similar protocol to the control group, but adherence to wearing offloading during weight-bearing activities is reinforced using a smartwatch. The smartwatch provides real-time reminders when participants walk without the offloading device. In addition, data from remote patient monitoring may help personalize education during weekly clinic visits conducted by the research coordinator.
  Interventions: Device: Offloading Boot

INTERVENTIONS:
Device: Offloading Boot — Removable offloading boot in one of three configurations provided to participants

SUMMARY:
The purpose of this study is to help people with diabetes who develop neuropathic diabetic foot ulcers (DFUs). These ulcers, or sores, if left untreated can increase the chance of amputation. Part of the treatment is to have the person wear a diabetic shoe or boot to help their foot heal. Sometimes people don't wear the boot like they are told. The investigators want to compare three different kinds of diabetic boots to see if they can help make it easier for people to wear their boots as instructed.

The investigators will look at three groups of participants: the first group will use removable offloading with reinforced education emphasizing continuous wear, including during rest and sleep, and not to remove it at any time. The second group will use removable offloading consistent with standard of care and receive education on recommended wear during walking or standing, with permission to remove the device during rest and sleep. The third group will use a smart removable offloading device that provides real-time adherence feedback via a smartwatch and smartphone, with additional personalized education informed by remotely monitored adherence data.

The investigators will also be looking at how much physical activity, like walking, the participants do. And they will compare how well participants sleep and rate their quality of life in the three different boots. The investigators think that giving participants information about how much they are wearing their boot using readily available technology will help them to follow the doctor's directions better, and help their wounds heal faster.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* ≥18 years old
* Non-infected, non-ischemic DFU requiring offloading
* Ambulatory at home with or without assistance
* Willing and able to provide written informed consent

Exclusion Criteria:

* Wound present for > 1 year
* HbA1c > 12%
* ABI of index limb < 0.6 or non-detectable Doppler, and/or patient being considered for revascularization during the course of the study
* Acute Charcot neuropathy or a major foot deformity that doesn't allow them to wear the smart boot
* Amputation proximal to the rearfoot on the affected extremity
* Any clinically significant medical or psychiatric condition
* Laboratory abnormality that would interfere with the ability to participate in the study
* Concurrently participating in exercise training
* Changes in psychotropic or sleep medication in the last 6 weeks
* Ulcer involves bone
* Ulcer not of diabetic origin
* Unable or unwilling to attend prescribed clinic visits or comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Wound healing at 12 weeks or sooner | Up to 12 weeks
  Wound healing is defined as complete epithelialization of the target ulcer, confirmed by standardized wound assessment. Healing status is recorded as a binary outcome (yes/no) for each participant. The proportion of participants achieving wound healing by 12 weeks is compared between randomized treatment arms.
  Unit of Measure: %
Time to wound healing | Up to 12 weeks
  Time to wound healing is defined as the number of days from randomization to confirm complete epithelialization of the target ulcer, as determined by standardized wound assessment.
  Unit of Measure: Days

SECONDARY OUTCOMES:
Patient acceptability | Week 12
  To evaluate participant acceptance of SmartBoot, the Technology Acceptance Model (TAM) questionnaire is administered. TAM is an intention-based framework widely used to assess user satisfaction and acceptance of new technologies. The questionnaire has 18 items: 9 assess perceived ease of use, 5 evaluate perceived benefits, 2 measure attitudes toward use, and 2 measure behavioral intention. Responses were rated on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). The average scores across all categories are normalized from 0 to 100; higher values indicate better acceptability. A score of 75 or higher is considered indicative of an acceptable level of program acceptance.
  Unit of Measure: unit on scale
Participant dropout rate | From baseline through Week 12
  Participant dropout is defined as discontinuation from the study before completion of the Week 12 visit. The dropout rate is calculated as the percentage of randomized participants who withdrew before Week 12.
  Unit of Measure: %
Adherence to offloading | From baseline through Week 12 (summarized weekly)
  The average weekly adherence to offloading is assessed using a SmartBoot adherence algorithm based on device-on time during weight-bearing activity or the patient's self-reports. The algorithm reports a normalized adherence score ranging from 1 to 10, with lower scores indicating better adherence to prescribed offloading and higher scores indicating poorer adherence.
  Unit of Measure: Unitless (normalized score, 1-10)
Percentage of Wound Area Reduction | Percent reduction in wound area per week
  The percentage of wound area reduction healing will be defined as the percentage reduction in wound area relative to baseline and estimated over time using a longitudinal linear model. Wound area will be derived from standardized wound imaging acquired weekly. When weekly wound area measurements are missing, values will be estimated using linear interpolation. Absolute wound area values (cm²) will also be retained in the database for descriptive purposes.
  - Unit of Measure: Percent reduction in wound area per week

OTHER OUTCOMES:
Change in gait speed | Baseline and monthly up to 12 weeks or until complete wound healing, whichever occurs first
  Gait speed (m/s) is assessed using validated wearable sensor-based measurements. Change in gait speed from baseline is calculated as the average change from baseline at each monthly follow-up assessment. A higher reduction indicates slower gait and potentially a sign of lower extremity muscle atrophy in response to offloading treatment.
  - Unit of Measure: m/s
Change in body sway area | Baseline and monthly up to 12 weeks or until complete wound healing, whichever occurs first
  * Outcome Measure Description: Postural control is assessed using validated wearable sensor-based measurements of body sway area (cm2) during quiet standing in a double-stance, eyes-open condition. Change in body sway area is calculated as the average change from baseline at each monthly follow-up assessment. A higher value can potentially be a sign of lower extremity muscle atrophy in response to offloading treatment.
  * Unit of Measure: cm^2
Sleep Quality | Baseline and monthly up to 12 weeks or until complete wound healing, whichever occurs first
  Sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI), which yields a global score ranging from 0 to 21, with higher scores indicating worse sleep quality. Scores greater than 5 have been used to indicate poor sleep quality and are reported here for descriptive interpretation.
  Unit of Measure: Unit on scale (0-21)
Overall Health | Baseline and monthly up to 12 weeks or until complete wound healing, whichever occurs first
  Overall health is assessed using the PROMIS-29 Profile, which measures seven health domains (Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles/Activities, and Pain Interference). Results are reported as T-scores standardized to the U.S. general population (mean = 50, SD = 10). For Physical Function and Social Roles, higher scores indicate better health; for all other domains, higher scores indicate greater symptom burden. Scores of 60 or higher on symptom scales or 40 or lower on function scales reflect moderate-to-severe impairment and are reported descriptively.
  Unit of Measure: T-score for each of 7 domains
Frailty (Trauma-Specific Frailty Index) | Baseline and monthly up to 12 weeks or until complete wound healing, whichever occurs first
  Frailty is assessed using the Trauma-Specific Frailty Index, calculated as the proportion of accumulated health deficits, with scores ranging from 0 to 1. Higher values indicate greater frailty. A value of approximately 0.25 will be used as a reference threshold for frailty and is reported descriptively.
  Unit of Measure: Unit on scale (0-1)
Frailty (Fried Frailty Criteria) | Baseline and monthly up to 12 weeks or until complete wound healing, whichever occurs first
  Frailty status is assessed using the Fried Frailty Criteria, which classify individuals based on five components. Scores range from 0 to 5, with higher scores indicating greater frailty. Categories of robust (0), pre-frail (1-2), and frail (≥3) are reported descriptively.
  Unit of Measure: Unit on scale (0-5)
Depressive symptoms | Baseline and monthly up to 12 weeks or until complete wound healing, whichever occurs first
  Depressive symptoms were assessed using the Center for Epidemiologic Studies Depression Scale (CES-D), which yields scores ranging from 0 to 60, with higher scores indicating greater symptom burden. Scores of 16 or higher will be used to indicate elevated depressive symptoms and are reported for descriptive purposes.
  Unit of Measure: Unit on scale (0-60)
Mobility Assessment | Baseline and monthly up to 12 weeks or until complete wound healing, whichever occurs first
  Mobility is assessed using the Life-Space Questionnaire, which yields scores ranging from 0 to 120, with higher scores indicating greater mobility. Lower scores reflect more restricted life-space mobility and are reported descriptively. Scores of 60 or lower are considered restricted life-space mobility.
  Unit of Measure: Unit on scale (0-120)
Fall Efficacy Score | Baseline and monthly up to 12 weeks or until complete wound healing, whichever occurs first
  Fear of falling is assessed using the Falls Efficacy Scale-International (FES-I), which yields scores ranging from 16 to 64, with higher scores indicating greater concern about falling. Scores of 28 or higher will be used to reflect a high concern about falling and are reported descriptively.
  Unit of Measure: Unit on scale (16-64)

CONTACTS AND LOCATIONS:
Overall Officials: David G Armstrong, DPN, MD, PhD, Principal Investigator — Professor of Surgery, Keck School of Medicine of USC
Locations (4):
- United States (4):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Verdugo Hills Hospital of USC, Glendale, California
  - Clemente Clinical Research, Los Angeles, California
  - Keck Medical Center of USC, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
Individually identifiable data will be deleted or masked before being made available to individuals who are not a part of the study (research staff). Results released will be sufficiently aggregated as to make individual identification of subjects highly unlikely. When individual research subjects are identifiable using substitute unique identifiers (i.e., subject 10) the translation table will be safeguarded from release outside of the study staff.
Supporting Information: Study Protocol, SAP